CLINICAL TRIAL: NCT06725407
Title: The Effects of Maternal Body Temperature Levels on Postoperative Maternal and Neonatal Results: a Cross-Sectional Study
Brief Title: Maternal Body Temperature in Caesarean Section
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sena Dilek Aksoy, Principal Investigator, Kocaeli University
Other Study IDs: sdilek11
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2021-01

CONDITIONS: Body Temperature Regulation
Keywords: Cesarean section; Birth; Body Temperature Regulation; Maternal Health; Newborn Health
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Cesarean section
  Interventions: Behavioral: Cesarean section

INTERVENTIONS:
Behavioral: Cesarean section — In the study, the participants' postoperative hypothermia development status was monitored.

SUMMARY:
The effect of maternal body temperature on the postpartum process and the newborn in innatal cesarean section is an important issue that needs to be emphasized. Hypothermia is defined as the patient's body temperature falling below 36.0 °C. Because hypothermia and shivering are frequently undesirable morbidities that occur during cesarean section. It can lead to many problems such as coagulopathy, increased transfusion requirement, surgical site infection, delayed metabolism of drugs, prolonged recovery, shivering and thermal discomfort. Many randomized controlled studies have been conducted on the heat regulation processes of women who gave birth by cesarean section, and maternal shivering and infection have been compared with parameters such as neonatal Apgar, blood pH and hypothermia. However, it is observational; data on care, breastfeeding, maternal mobilization and comfort are limited. The aim of this study was to determine the postoperative maternal and neonatal effects of maternal body temperature after cesarean section. An analytical cross-sectional study design will be used. All samples meeting the inclusion criteria of the study will be reached between 10.01.2021-10.01.2022. Research data will be collected using the pregnancy information form, postoperative maternal-neonatal follow-up form, Facial Pain Scale and Temperature Comfort Perception Scale. Research data will be collected using the IBM SPSS Statistic program.

DETAILED DESCRIPTION:
Research questions

1. What is the prevalence of maternal hypothermia in women who deliver by cesarean section?
2. What are the effects of maternal hypothermia on postoperative maternal vital signs, pain, mobilization, nutrition, digestive system, thermal comfort, and breastfeeding in women who deliver by cesarean section?
3. What are the effects of maternal hypothermia on neonatal vital signs, Apgar score, first sucking activity, nutrition, oxygen, and intensive care unit requirements in women who deliver by cesarean section? The study will be conducted with an analytical cross-sectional design. The study population will consist of women who gave birth by planned cesarean section in a state hospital in Turkey between 10.01.2021 and 10.01.2022.

The data of the study will be collected using the Pregnant Women Information Form, Postoperative Maternal and Neonatal Follow-up Forms, Faces Pain Scale (FPS) and Thermal Comfort Perception Scale (TCPS).

Statistical analyzes of the data will be performed using IBM SPSS (IBM Corp., NY, USA). Descriptive statistics (number, percentage, mean, standard deviation) will be used to evaluate sociodemographic data. In the comparison of categorical variables, parametric tests (Chi-square, t test, etc.) will be used when the data are normally distributed, and nonparametric tests (Mann-Whitney U test, Kruskal-Walli test, etc.) and regression analysis will be used when the data are not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 18 years of age or older,
* Able to answer the research questions,
* Without any contagious disease including middle ear infection,
* Volunteer

Exclusion Criteria:

* Those with clotting disorders,
* Thyroid disease,
* Those with a body mass index below 18.5,
* Those with mental problems that prevent them from answering questions,
* Those whose babies were born with anomalies,
* Those who had a stillbirth,
* Those who were given special heated blankets and fluids

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women between the ages of 18-45 who have been given the decision to have a planned caesarean section.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Postoperative hypothermia | Postoperative Day 0 (will be measured at 1st hour, 6th hour, 12th hour and 24th hour)

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Associate Professor, Ph.D., Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No